CLINICAL TRIAL: NCT05966233
Title: Phase II Randomized Clinical Trial to Evaluate the Efficacy of the Addition of Polatuzumab Vedotin to Standard Chemotherapy R-DHAP (POLA-R-DHAP) as Induction Pre-transplantation Therapy in Patients With Diffuse Large B-Cell Lymphoma Refractory/Relapsed After First Line Treatment.
Brief Title: R-DHAP vs POLA-R-DHAP Followed by Autologous Transplant as First Salvage Treatment in Patient With Relapsed or Refractory Diffuse Large B Cell Lymphoma
Acronym: FIL_POLARDHAP
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIL_POLA-R-DHAP
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Diffuse Large B Cell Lymphoma Refractory; Diffuse Large B-cell Lymphoma Recurrent
Keywords: Lymphoma; Diffuse Large B cell Lymphoma; Immunochemotherapy; DLBCL; Autologous; Transplant; Relapsed; Refractory; DHAP; Rituximab; Polatuzumab Vedotin; Randomized; R-DHAP; CD79; PET; Review
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R-DHAP (Active Comparator): R-DHAP x4 + autologous transplant/salvage treatment (based on centrally review response)
  Interventions: Drug: R-DHAP
- Pola-R-DHAP (Experimental): Pola-R-DHAP x4 + autologous transplant/salvage treatment (based on centrally review response)
  Interventions: Drug: Pola-R-DHAP

INTERVENTIONS:
Drug: R-DHAP — * Rituximab 375 mg/m2 IV on D0 or D1
  * Dexamethasone 40 mg/day IV or PO on D1-4
  * Ara-C 2 g/m2 IV on D2 (2 doses every 12h) or D2 and D3
  * Cisplatin 100 mg/ m2 IV on D1
  Arms: R-DHAP
Drug: Pola-R-DHAP — * Polatuzumab Vedotin 1.8 mg/kg IV on D1
  * Rituximab 375 mg/m2 IV on D0 or D1
  * Dexamethasone 40 mg/day IV or PO on D1-4
  * Ara-C 2 g/m2 IV on D2 (2 doses every 12h) or D2 and D3
  * Cisplatin 100 mg/ m2 IV on D1
  Arms: Pola-R-DHAP

SUMMARY:
Prospective, multicenter, open label, phase II randomized clinical trial in DLBCL patients relapsed or refractory to first line R-chemo, aged 18-70 years and candidate to autologous transplant. Patients will be randomized 1:1 to received 4 cycles of R-DHAP or R-DHAP plus Polatuzumab Vedotin as induction treatment plus autologous transplant.

DETAILED DESCRIPTION:
Prospective, multicenter, open label, phase II randomized clinical trial in DLBCL patients relapsed or refractory to first line R-chemo, aged 18-70 years and candidate to autologous transplant. Patients will be randomized 1:1 to received 4 cycles of R-DHAP or R-DHAP plus Polatuzumab Vedotin as induction treatment.

PET-CT scan performed after induction be centrally review for disease response. Responding patients (CR) after induction will be addressed to receive Autologous Stem Cells Transplantation (ASCT) consolidation as per local guidelines. Patients achieving PR can proceed with ASCT or with a 3rd-line treatment, according to the physician judgment. Patients in SD/PD will be diverted to salvage strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented diagnosis of Diffuse Large B-Cell Lymphoma Not otherwise specified (DLBCL-NOS) as defined in the 2022 edition of the World Health Organization (WHO) classification; are also admitted documented diagnosis of:

   * T-cell/histiocyte-rich large B-cell lymphoma (THRLBCL)
   * Epstein-barr virus (EBV)-associated DLBCL
   * Double-hit and triple-hit high grade B-cell lymphomas (HGBL DH/TH)
   * High-grade B-cell lymphoma, NOS (HGBL)
   * Transformed FL not previously untreated
   * Follicular large B-cell lymphoma (FLBL, former follicular 3b)
2. Known availability of biopsy material (at relapse/refractory or previous most recent). Re-biopsy highly encouraged even if not mandatory. Central pathology review required, but not mandatory for registration and treatment start;
3. Relapse or refractoriness after the first line R-chemo (R-CHOP o similar). Previous treatment with polatuzumab containing regimen is allowed as per clinician judgment;
4. CAR-T not indicated or unavailable;
5. Age 18-70 years. sGA mandatory for patients 65-70 years old: only category FIT admitted [20] (see Appendix A);
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 if not related to lymphoma disease (see Appendix B);
7. Measurable disease ≥ 1.5 cm in longest diameter, and measurable in 2 perpendicular dimensions;
8. Normal blood count defined as: neutrophils at least 1.500/mmc, platelets at least 75.000/mmc, haemoglobin at least 8,0 g/dL with transfusion independence, unless abnormalities due to underlying disease (bone marrow involvement), at the moment of signing informed consent;
9. Adequate liver function, assessed by baseline laboratory values; the increase to up to 2.5 ULN for transaminases and up to 1.5 ULN for bilirubin admitted for cases with documented liver involvement by lymphoma;
10. Adequate renal function defined as creatinine clearance ≥ 40 mL/min (Cockcroft-Gault formula; see Appendix C)
11. Subjects HBsAg negative but positive for antibodies to hepatitis B core antigen with undetectable HBV-DNA measured by real-time polymerase chain reaction (PCR).
12. Women of childbearing potential (WOCBP) and men must agree to use effective contraception if sexually active. Females of childbearing potential and males with female partners of reproductive potential should be advised to use effective contraception while receiving polatuzumab vedotin and for 9 months after the last dose of polatuzumab vedotin for female patients and for 6 months after the last dose of polatuzumab vedotin for male patients with female partners of reproductive potential. A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include but are not limited to hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for continuous 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. The investigator or a designated associate is requested to advise the patient how to achieve highly effective birth control method (failure rate of less than 1%) e.g. intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner. The use of condoms by male patients is required (even if surgically sterilized, i.e., status post vasectomy) unless the female partner is permanently sterile. Full sexual abstinence is admitted when this is in line with the preferred and usual lifestyle of the subject, for the same time period planned for other methods of birth control (see above). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods for the female partner) and withdrawal are not acceptable methods of contraception
13. WOCBP must have a negative serum (beta-human chorionic gonadotropin [b-hCG]) or urine pregnancy test at Screening. Women who are pregnant or breastfeeding are ineligible for this study;
14. Life expectancy > 6 months;
15. Subject understands and voluntarily signs an informed consent form approved by the National Ethics Committee prior to the initiation of any screening or study-specific procedures;
16. Subject must be able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Any histology other than DLBCL
2. Primary mediastinal lymphoma (PMBCL)
3. Known central nervous system lymphoma
4. Known history of severe allergic or anaphylactic reactions to human, humanized, chimeric, or murine monoclonal antibodies
5. Contraindication to any drug in the chemotherapy regimen
6. Left ventricular ejection fraction (LVEF) < 50%
7. Neuropathy ≥ grade 2
8. Subject is:

   * Seropositive for hepatitis B, defined by a positive test for hepatitis B surface antigen [HBsAg]. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (HBsAb positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR
   * Known to be seropositive for hepatitis C. EXCEPTION: Patients with presence of HCV antibody, but PCR negative for HCV-RNA are eligible
   * Positive for human immunodeficiency virus (HIV) infection
9. Any uncontrolled active systemic infection requiring intravenous (IV) antibiotics
10. History of stroke or intracranial hemorrhage within the past 6 months.
11. History of clinically relevant liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, rheumatologic, hematologic, psychiatric, or metabolic disturbances
12. Clinically significant cardiovascular disease
13. Major surgical intervention prior 4 weeks to enrollment if not due to lymphoma and/or other disease life-threatening that can compromise chemotherapy treatment
14. Prior malignancies other than lymphoma in the last 5 years with exception of currently treated basal or squamous cell carcinoma or melanoma of the skin or in situ carcinoma of the cervix
15. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety
16. If female, the patient is pregnant or breast-feeding
17. Patients participating in other clinical studies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From treatment start up to 30 months (6 months treatment period and 24 months of follow-up)
  Time between the randomization to first documentation of recurrence, progression or death from any cause

SECONDARY OUTCOMES:
Event-Free Survival (EFS) | From treatment start up to 30 months (6 months treatment period and 24 months of follow-up)
  Time between the randomization to any treatment failure, including disease progression, or discontinuation of treatment for any reason (e.g., disease progression, toxicity, patient preference, initiation of a new treatment without documented progression) or death from any cause.
Complete response rate (CRR) | From treatment start up to end of treatment evaluation (about 6 months)
  CRR will be defined according to Response Criteria for NHL with PET (Lugano 2014). CRR will include only patients who achieved a CR and will be evaluated on assessed patients and on all treated patients, considering patients without a response assessment (due to any reason) as non-responders.
Overall response rate (ORR) | From treatment start up to end of treatment evaluation (about 6 months)
  ORR will be defined as the proportion of patients who have a partial or complete response to therapy (CR+PR).
Overall Survival (OS) | From treatment start up to 30 months (6 months treatment period and 24 months of follow-up)
  Time between randomization to death from any cause.
Incidence and severity of AEs | From start to end of induction treatment evaluation (about 3 months)
  Incidence and severity of AEs in R-DHAP vs POLA-R-DHAP according to latest CTCAE criteria during induction immunochemotherapy
Adequate stem cells mobilization | From beginning of 2nd cycle to end of induction treatment evaluation (about 2 months)
  Adequate stem cells mobilization will be defined by the target cell harvesting of 3 x 10^6 CD34+ cells/kg
Autologous consolidation feasibility | At time of end of treatment assessment (up to 6 months from treatment begin)
  Proportion of patients receiving autologous consolidation after POLA-R-DHAP vs R-DHAP

CONTACTS AND LOCATIONS:
Overall Officials: Monica Balzarotti, MD, Principal Investigator — Dipartimento di Oncologia Medica ed Ematologia - Istituto Clinico Humanitas - Rozzano (MI)
Locations (37):
- Italy (37):
  - A.O. SS. Antonio e Biagio e Cesare Arrigo, S.C. Ematologia, Alessandria
  - AOU Ospedali Riuniti, Clinica di Ematologia, Ancona
  - Azienda Ospedaliera S.Giuseppe Moscati, S.C. Ematologia e Trapianto emopoietico, Avellino
  - IRCCS Centro di Riferimento Oncologico di Aviano, Divisione di Oncologia e dei Tumori immuto-correlati, Aviano
  - IRCCS Istituto Tumori Giovanni Paolo II, U.O.C Ematologia, Bari
  - Cliniche Humanitas Gavazzeni, Oncologia, Bergamo
  - ASST Spedali Civili di Brescia, Ematologia, Brescia
  - Fondazione del Piemonte per l'Oncologia - IRCCS, Ematologia, Candiolo
  - Arnas Nuovo Ospedale Garibaldi Nesima, U.O.C. Ematologia, Catania
  - A.O. S. Croce e Carle, S.C. di Ematologia e Trapianto di Midollo Osseo, Cuneo
  - Azienda Ospedaliera Universitaria Careggi, Unitа funzionale di Ematologia, Florence
  - Ospedale Vito Fazzi, Ematologia, Lecce
  - ASST Ovest Milanese - Legnano, U.O.C. Ematologia, Legnano
  - ASST Grande Ospedale Metropolitano Niguarda, SC Ematologia, Milan
  - Istituto Scientifico San Raffaele, Unitа Linfomi - Dipartimento Oncoematologia, Milan
  - Ospedale Maggiore Policlinico - Fondazione IRCCS Ca Granda, Ematologia, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Ematologia, Monza
  - AOU Maggiore della Caritа di Novara, SCDU Ematologia, Novara
  - A.O. Ospedali Riuniti Villa Sofia-Cervello, Divisione di Ematologia, Palermo
  - Ospedale S. Maria della Misericordia, Ematologia, Perugia
  - P.O. Spirito Santo di Pescara, UOS Dipartimentale - Centro di diagnosi e Terapia dei linfomi, Pescara
  - Ospedale Guglielmo da Saliceto, U.O.Ematologia, Piacenza
  - AOU Pisana, U.O. Ematologia, Pisa
  - A.O.R. "San Carlo", U.O. Ematologia, Potenza
  - Ospedale delle Croci, Ematologia, Ravenna
  - Azienda Unitа Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova, Ematologia, Reggio Emilia
  - AO San Giovanni Addolorata, S.C. Ematologia, Roma
  - AO Sant Andrea, Ematologia, Roma
  - Policlinico Umberto I - Universitа "La Sapienza", Istituto Ematologia -Dipartimento di Medicina Traslazionale e di Precisione, Roma
  - Policlinico Universitario Campus Bio-Medico, Ematologia - Trapianto cellule staminali - Medicina Trasfusionale e Terapia cellulare, Roma
  - Istituto Clinico Humanitas, U.O. Ematologia, Rozzano
  - AOU Senese, U.O.C. Ematologia, Siena
  - A.O.U. Citta della Salute e della Scienza di Torino, Ematologia Universitaria, Torino
  - A.O.U. Citta della Salute e della Scienza di Torino, S.C.Ematologia, Torino
  - Ospedale Ca Foncello, S.C di Ematologia, Treviso
  - A.O.C. Panico, U.O.C Ematologia e Trapianto, Tricase
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI), SC Ematologia, Trieste